CLINICAL TRIAL: NCT02541890
Title: Effects of Workplace Intervention in Inpatient Occupational Rehabilitation on Return to Work for Persons With Somatic and/or Common Mental Health Problems. A Randomised Controlled Trial
Brief Title: Effects of Workplace Intervention in Occupational Rehabilitation on Return to Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Trondheim University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/2279
Record Dates: First submitted 2015-08-18; First posted 2015-09-04 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Mental Disorders; Musculoskeletal Diseases; Fatigue Syndrome, Chronic
Keywords: Rehabilitation; Return to Work
MeSH Terms: conditions — Mental Disorders; Musculoskeletal Diseases; Fatigue Syndrome, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Work place intervention (Experimental): Work place intervention in addition to rehabilitation program.
  Interventions: Behavioral: Work place intervention
- Rehabilitation program only (No Intervention): Rehabilitation program without intervention at the work place.

INTERVENTIONS:
Behavioral: Work place intervention — Meeting at the work place including the patient, the employer and the rehabilitation therapist. Aim of meeting is to discuss challenges and possibilities in the patient's return to work process and to make a plan for return to work.
  Arms: Work place intervention

SUMMARY:
Aim is to study the effect of a work place intervention during a multicomponent return-to-work rehabilitation program on return-to-work. The intervention is compared with inpatient rehabilitation only, and participants will be recruited from the diagnostic groups dominating the sick-leave statistics, namely musculoskeletal disorders, common mental disorders (e.g. stress, depression and anxiety), and unspecific disorders including chronic fatigue.

DETAILED DESCRIPTION:
Long-term sick-listing from work has considerable impact on social function, on the families of the sick-listed persons, the companies they work for, and society as a whole. Hence, the need for documented effective vocational rehabilitation programs is pressing. Vocational rehabilitation services described in the scientific literature have been specific to one single or a specific group of medical conditions (e.g.low back pain). In contrast, most people on sick leave have several health complaints, and many of the factors influencing sick leave are shared regardless of disorder (e.g. social surroundings, workplace environment), calling for rehabilitation programs that can be employed for both musculoskeletal, unspecific and common mental disorders. Research indicates that interventions on the work place might facilitate return to work. The aim of this study is therefore to investigate the effect of a work place intervention during a multicomponent return-to-work rehabilitation program on return-to-work.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Central Norway
* Sick-listed due to common mental disorders, musculoskeletal pain/problems, unspecific disorders and/or fatigue
* Sick-listed more than 50 %
* Sick-listed longer than 8 weeks
* Has employer and is willing to participate in a work place intervention during the rehabilitation program

Exclusion Criteria:

* is self-employed
* has, or is currently examined for, a serious somatic or psychiatric disorder
* suffers from substance abuse
* has trouble with participating in a group
* is in a rehabilitation process that will interfere with the occupational rehabilitation program
* function level is to weak to participate in the rehabilitation program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of days on sick-leave | 12 months
  Register data from the national health and welfare services
Time until sustainable return to work | 12 months
  Register data from the national health and welfare services

SECONDARY OUTCOMES:
Use of health services. Questionnaire. "How much of this health/social service have you used during the last 4 months?" | 12 months
  160 participants. "How much of this health/social service have you used during the last 4 months?" Somatic and mental health specialized care (in-patient and outpatient), general practitioner, psychologist, group therapy, physiotherapist, chiropractor, occupational rehabilitation, welfare services, complementary practitioner, emergency unit, ambulatory services, occupational health services, other treatment.
Pain. Questionnaire | 12 months
  Brief pain inventory (BPI). 160 participants
Health related quality of life. Questionnaire | 12 months
  The 15D health-related quality of life instrument. 160 participants
Psychological flexibility and acceptance. Questionnaire | 5 months
  Acceptance and action questionnaire and work acceptance and action questionnaire (AAQ2). 160 participants
Return to work self efficacy. Questionnaire. | 5 months
  Return to work self-efficacy-19 (RTWSE-19). 160 participants.
Fear and avoidance beliefs about work. Questionnaire | 5 months
  Fear Avoidance Belief Questionnaire (FABQ). 160 participants
Expectations about sick leave and return to work. Questionnaire | 5 months
  160 participants. "How long do you anticipate to be sick-listed (partly/fully)?" 3 questions.
Work ability. Single question | 5 months
  160 participants. "How will you rate your work ability?" (scale from 0 (no ability) to 10 (my best ability)).
Well-being at work. Single question | 5 months
  160 participants. "How happy are you at work?" (not at all, not so good, good. very good)
Readiness for return to work. Questionnaire | 5 months
  160 participants. Readiness for return to work (RRTW) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marius S Fimland, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Nowegian University of Science and Technology, Department of public health, Trondheim, Norway

REFERENCES:
- [Background] Rise MB, Skagseth M, Klevanger NE, Aasdahl L, Borchgrevink P, Jensen C, Tenggren H, Halsteinli V, Jacobsen TN, Loland SB, Johnsen R, Fimland MS. Design of a study evaluating the effects, health economics, and stakeholder perspectives of a multi-component occupational rehabilitation program with an added workplace intervention - a study protocol. BMC Public Health. 2018 Feb 5;18(1):219. doi: 10.1186/s12889-018-5130-5. PMID 29402253
- [Result] Skagseth M, Fimland MS, Rise MB, Johnsen R, Borchgrevink PC, Aasdahl L. Effectiveness of adding a workplace intervention to an inpatient multimodal occupational rehabilitation program: A randomized clinical trial. Scand J Work Environ Health. 2020 Jul 1;46(4):356-363. doi: 10.5271/sjweh.3873. Epub 2019 Dec 13. PMID 31834410
- [Result] Klevanger NE, Fimland MS, Rise MB. Aligning stakeholders' understandings of the return-to-work process: a qualitative study on workplace meetings in inpatient multimodal occupational rehabilitation. Int J Qual Stud Health Well-being. 2021 Dec;16(1):1946927. doi: 10.1080/17482631.2021.1946927. PMID 34278973